CLINICAL TRIAL: NCT01366079
Title: Dynamic Position Change in Colonic Adenoma Detection: a Prospective, Randomized, Multicenter Study
Brief Title: Dynamic Position Change in Colonic Adenoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong-Seon Ji, MD, PhD, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dynamic study
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Position; Colonoscopy; Adenoma
MeSH Terms: conditions — Adenoma

ARMS (2):
- Position change (Experimental): Position change group
  Interventions: Procedure: Position change
- Left lateral (Active Comparator): Left lateral position
  Interventions: Procedure: Left lateral

INTERVENTIONS:
Procedure: Position change — Patients change position (cecum to hepatic flexure, left lateral; transverse colon, supine; splenic flexure and descending colon , right lateral) during colonoscopy withdrawal.
  Arms: Position change
Procedure: Left lateral — In left lateral position group patients are positioned left lateral decubitus during colonoscopy withdrawal.
  Arms: Left lateral

SUMMARY:
There was an only single operator study reporting dynamic position change during colonoscopy withdrawal significantly improved polyp and adenoma detection. So we designed a prospective, randomized multicenter study to verify the effect of dynamic position change in colonic adenoma detection. We think position change improve luminal distension and has the potential to improve adenoma detection rate.

ELIGIBILITY:
Inclusion Criteria:

* patient aged over 45 years who will be performed colonoscopy for the first time

Exclusion Criteria:

* polyposis syndrome
* musculoskeletal problem
* Inflammatory bowel disease
* previous bowel operation

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Adenoma detection | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Korea, Incheon, Daejeon, Bucheon, Seoul, South Korea